CLINICAL TRIAL: NCT00848783
Title: A Randomized Phase-II Study of Patients With Locally Advanced Gastric of Gastro-Esophageal Adenocarcinoma Treated With Induction Irinotecan/Cisplatin, Potentially Curative Surgery With or Without Adjuvant Intraperitoneal Floxuridine, Followed by Prolonged Administration of Capecitabine
Brief Title: Irinotecan/Cisplatin, Potentially Curative Surgery With or Without Floxuridine, Followed by Capecitabine for Stomach and Gastro-esophageal Junction (GEJ) Cancers
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Due to slow accrual
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 07-837; NYU 05-20 (Other: NYU medical center)
Record Dates: First submitted 2009-02-19; First posted 2009-02-20 (Estimated); Results first posted 2012-12-10 (Estimated); Last update posted 2018-01-08 (Actual); Status verified 2017-12

CONDITIONS: Gastric Cancer; Gastric Adenocarcinoma; Esophageal Cancer
Keywords: gastric cancer; gastroesophageal junction; stomach cancer; intraperitoneal infusion; capecitabine; irinotecan; cisplatin; floxuridine
MeSH Terms: conditions — Stomach Neoplasms; Esophageal Neoplasms | interventions — Irinotecan; Cisplatin; Surgical Procedures, Operative; Floxuridine; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A-with IP Floxuridine (Experimental): 1. Induction treatment:
     Cisplatin 25 mg/m^2 and Irinotecan 75 mg/m^2 once a week for 4 weeks, both intravenous; Two weeks without treatment; Repeat the course once.
  2. Re-evaluation, surgery if complete response, partial response or stable disease, or off the protocol if progression of disease.
  3. Randomization
  4. Surgery.
  5. Postoperative IP treatment:
     Day 1,2,3: Floxuridine 3 gm/day, IP; Day 3: Cisplatin 60 mg/m^2, IP; 2 weeks without treatment; repeat the course once
  6. Postoperative systemic treatment: courses 1-9: Capecitabine 2,000 mg/m^2/day x14 every 3 weeks/course, Oral
  Interventions: Drug: Irinotecan; Drug: Cisplatin; Procedure: Surgery; Drug: Floxuridine; Drug: Capecitabine
- B-Without IP Floxuridine (Experimental): Same as Arm A except no postoperative IP treatment.
  Interventions: Drug: Irinotecan; Drug: Cisplatin; Procedure: Surgery; Drug: Capecitabine

INTERVENTIONS:
Drug: Irinotecan
  Other Names: CPT-11
Drug: Cisplatin
Procedure: Surgery
Drug: Floxuridine
  Other Names: FUDR
  Arms: A-with IP Floxuridine
Drug: Capecitabine
  Other Names: Xeloda

SUMMARY:
This study is to determine whether intraperitoneal (IP) Floxuridine is effective in the patients with advanced stomach or gastro-esophageal junction cancers in the treatment consisting of pre- and post-surgery chemotherapies.

DETAILED DESCRIPTION:
A previous Phase-II trial conducted by the same principle investigator(s), utilizing preoperative chemotherapy and intraperitoneal consolidation, was conducted in patients with locally advanced, potentially resectable gastric cancer or cancer of the gastro-esophageal junction (GEJ), both staged as T3N0, T4N0, any TN1 or TN2 disease. The data suggest that for patients with locally advanced gastric or GEJ cancer, systemic induction therapy, curative surgery with high Ro resection rates, and IP adjuvant therapy, has acceptable toxicity and encouraging survival outcome. The Medical Research Council Adjuvant Gastric Infusional Chemotherapy (MAGIC) trial has also shown that perioperative chemotherapy - chemotherapy given both before and after surgery - can provide a significant survival benefit.

The investigators hypothesize that adjuvant intraperitoneal salvage of cancer micrometastatic residues after surgery contributes to disease-free survival. The goal of this trial is to determine whether IP Floxuridine, added to adjuvant postoperative chemotherapy, prolongs patient's survival. This will be tested during the randomized open-label trial.

ELIGIBILITY:
* Only untreated patients with histologically documented gastric/GEJ adenocarcinoma, clinical American Joint Committee on Cancer (AJCC) stage grouping (11) IB-IV (Mo) by CT scan and laparoscopy/endoscopic ultrasound, are eligible. Excluded are patients in need of urgent surgery for gastro-intestinal obstruction, perforation or hemorrhage.
* Both men and women >= 18 years of age with Eastern Cooperative Oncology Group (ECOG) performance status 0-2, members of any ethnic group and minorities.
* Patients without another invasive malignancy, with adequately treated basal cell or squamous cell skin cancer, free for 5 years or more of in-situ cervix cancer or other in-situ cancer.
* Since immune deficiency increases the risk of terminal infections when aggravated by bone marrow suppressive therapy, patients must be without active or uncontrolled infection including HIV.
* Patients without psychiatric disorders that may interfere with their consent and/or with protocol follow-up.
* An adequate bone-marrow reserve (absolute neutrophil count >= 1,500/ mmL, thrombocytes >= 100,000 mmL, hemoglobin >= 9 gm/dL).
* Preserved liver and renal function (total serum bilirubin <2 mg/dL, SGOT/SGPT =< 3x the upper limit of normal, alkaline phosphatase =< 3x the upper limit of normal, blood urea nitrogen (BUN) =< 30 mg/dL, serum creatinine concentration <1.5 mg/dL and creatinine clearance >= 50 mL/min) are required. Creatinine clearance should be normalized for 1.73 M^2 BSA. The prothrombin time, activated partial thromboplastin time, and thrombin time should be within the range of normal values.
* Since chemotherapeutic agents to be used are known or suspected to be teratogenic or with other adverse effects, women must not be pregnant or breast-feeding. All females of childbearing potential must have a blood test or urine study within 2 weeks prior to registration to rule out pregnancy. All patients of reproductive age may not participate unless they agree to use an effective medically acceptable contraceptive method.
* Patients without diagnosed Gilbert's disease and bilirubin level >= 2.0 mg/dL, as these patients may have excessive CPT-11 toxicity.
* No prior severe reaction to fluoropyrimidine therapy or known hypersensitivity to 5-fluorouracil. Capecitabine (Xeloda) is contraindicated in patients with severe renal impairment, i.e., creatinine clearance below 30 mL/min, determined by Cockcroft-Gault equation shown on page 15 under (i) Renal impairment. In patients with moderate renal impairment (creatinine clearance 30-50 mL/min), which develops during the course of adjuvant treatment with Capecitabine, the drug is decreased to 75% of the starting dose.
* Patients should be without any severe concurrent disease, such as cardiac condition not responding to medication, myocardial infarction within the last 12 months, active infection or uncontrolled pulmonary disease, or any other disease which in judgment of the investigator would make the patient inappropriate for entry into this study.
* Patients who signed written informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2008-05; Primary Completion 2011-08 (Actual); Study Completion 2012-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Franco Muggia, MD, Principal Investigator — NYU Langone Health
Locations (3):
- United States (3):
  - Norris Cancer Center, Los Angeles, California
  - Bellevue Hospital, New York, New York
  - NYU Cancer Center, New York, New York

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between March 2008 and May 2010 eight patient were enrolled to the study from New York University Langone Medical Center and University of South California Cancer Center.
Pre-assignment Details: Patients were randomized to Arm A or Arm B after the response evaluation of the induction treatment. One patient was not randomized due to progression of disease before surgery and was taken off the protocol treatment.
Groups:
- Induction Treartment Only: This is not a treatment cohort specified in the protocol. The patient in this group was not randomized to Arm A or Arm B due to disease progression before surgery and was taken off the study.
Period: Overall Study
Arm/Group | A-with IP Floxuridine | B-Without IP Floxuridine | Induction Treartment Only
Started | 4 | 3 | 1
Completed | 1 | 1 | 1
Not Completed | 3 | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Induction Treatment Only: This is not a treatment cohort specified in the protocol. The patient in this group was not randomized to Arm A or Arm B due to disease progression before surgery and was taken off the study.
- Total: Total of all reporting groups
Arm/Group | A-with IP Floxuridine | B-Without IP Floxuridine | Induction Treatment Only | Total
Number analyzed (Participants) | 4 | 3 | 1 | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 4 | 3 | 1 | 8
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.8 (12.8) | 54.3 (3.2) | 60 (0) | 54.8 (8.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 0 | 1
  Male | 3 | 3 | 1 | 7
Region of Enrollment [Number; unit: participants]
  United States | 4 | 3 | 1 | 8

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With One-year Recurrence-free Survival
Description: This is defined as the patients who did not have recurrence of cancer at 1 year since the start of induction chemotherapy.
Time Frame: 1 year
Population: Based on intent-to-treat population.
Measure: Number; unit: participants
Arm/Group | A-with IP Floxuridine | B-Without IP Floxuridine
Number analyzed (Participants) | 4 | 3
participants | 3 | 2

2. Secondary Outcome: Overall Survival Rate; Toxicity; Evaluation of Sites of Relapse of Failing Patients
Description: Secondary outcome measure was not analyzed as study was terminated
Time Frame: every 4 months for the first 2 years, every 6 months for years 3 and 4, then every 12 months for up to 10 years
Population: Secondary outcome measure was not analyzed as study was terminated
Arm/Group | A-with IP Floxuridine | B-Without IP Floxuridine | Induction Treatment Only
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: The adverse events were followed during the whole treatment phase, about 1 year.
Arm/Group | A-with IP Floxuridine | B-Without IP Floxuridine
Serious Adverse Events (participants affected / at risk) | 0/4 | 2/3
Other Adverse Events (participants affected / at risk) | 4/4 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | A-with IP Floxuridine (N=4) | B-Without IP Floxuridine (N=3)
Neutrophils/Granulocytes (Anc/Agc) (Blood and lymphatic system disorders) | 0 | 1
Infection With Normal Anc Or Grade 1 Or 2 Neutrophils (Infections and infestations) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | A-with IP Floxuridine (N=4) | B-Without IP Floxuridine (N=3)
Blood/Bone Marrow - Other (Specify, __) (Blood and lymphatic system disorders) | 1 | 0
Hemoglobin (Blood and lymphatic system disorders) | 4 | 1
Palpitations (Cardiac disorders) | 1 | 0
Fatigue (Asthenia, Lethargy, Malaise) (General disorders) | 4 | 1
Insomnia (General disorders) | 2 | 0
Weight Loss (General disorders) | 2 | 0
Hair Loss/Alopecia (Scalp Or Body) (Skin and subcutaneous tissue disorders) | 2 | 0
Anorexia (Gastrointestinal disorders) | 2 | 1
Constipation (Gastrointestinal disorders) | 2 | 0
Diarrhea (Gastrointestinal disorders) | 4 | 2
Distension/Bloating, Abdominal (Gastrointestinal disorders) | 2 | 0
Dysphagia (Difficulty Swallowing) (Gastrointestinal disorders) | 1 | 0
Heartburn/Dyspepsia (Gastrointestinal disorders) | 1 | 1
Nausea (General disorders) | 4 | 1
Taste Alteration (Dysgeusia) (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 3 | 1
Alt, Sgpt (Serum Glutamic Pyruvic Transaminase) (Investigations) | 1 | 0
Ast, Sgot(Serum Glutamic Oxaloacetic Transaminase) (Investigations) | 1 | 0
Glucose, Serum-High (Hyperglycemia) (Metabolism and nutrition disorders) | 2 | 0
Dizziness (Nervous system disorders) | 2 | 0
Mood Alteration (Nervous system disorders) | 1 | 0
Neurology - Other (Specify, __) (Nervous system disorders) | 2 | 0
Neuropathy: Sensory (Nervous system disorders) | 1 | 1
Pain (General disorders) | 3 | 0
Neutrophils/Granulocytes (Anc/Agc) (Blood and lymphatic system disorders) | 3 | 1
Platelets (Blood and lymphatic system disorders) | 1 | 0

LIMITATIONS AND CAVEATS:
Early termination leading to small numbers of subjects analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No